CLINICAL TRIAL: NCT04008992
Title: A Randomized, Double-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of BMS-986259 in Healthy Participants.
Brief Title: An Ascending Dose Study of BMS-986259 to Study Safety in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CV019-002
Record Dates: First submitted 2019-06-20; First posted 2019-07-05 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part A SAD - A1 Cohort (Experimental): Single Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part A SAD - A2 Cohort (Experimental): Single Ascending dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part A SAD- A3 Cohort (Experimental): Single Ascending dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part A SAD- A4 Cohort (Experimental): Single Ascending dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part A SAD - A5 Cohort (Experimental): Single Ascending dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part A SAD- A6 Cohort (Experimental): Single Ascending dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part B MAD- B1 Cohort (Experimental): Multiple Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part B MAD - B2 Cohort (Experimental): Multiple Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part B MAD - B3 Cohort (Experimental): Multiple Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part B MAD - B4 Cohort (Experimental): Multiple Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part C JMAD - C1 Cohort (Experimental): Japanese Multiple Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part C JMAD - C2 Cohort (Experimental): Japanese Multiple Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol
- Part C JMAD - C3 Cohort (Experimental): Japanese Multiple Ascending Dose
  Interventions: Drug: BMS-986259; Other: Placebo; Diagnostic Test: P-Aminohippurate; Diagnostic Test: Iohexol

INTERVENTIONS:
Drug: BMS-986259 — Single and Multiple ascending dose from Dose 1 to Dose 5
Other: Placebo — Placebo matching BMS-986259
Diagnostic Test: P-Aminohippurate — Diagnostic Agent
Diagnostic Test: Iohexol — Diagnostic Agent

SUMMARY:
A Randomized double blind, placebo controlled study of BMS-986259 to evaluate the safety and effectiveness of the drug amongst different conditions and populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with a body mass Index (BMI) of 18.0 kg/m^2 - 30.0 kg/m^2.
* Males and females not of child bearing potential.
* Participants in the Japanese Cohorts in Part C must be first-generation Japanese (born in Japan, not living outside of Japan for more than 10 years, and both parents are ethnically Japanese.)

Exclusion Criteria:

* Any previous dosing in another cohort in the current study or participation in an investigational drug within 2 months prior to (the first) drug administration in the current study.
* Any Significant Acute or Chronic medical Illness, major surgery in 12 months, or so smoking or used smoking cessation in 3 months.
* Inability to be venipunctured and/or tolerate venous access. ,abnormalities in hemoglobin or positive screen for hepatitis C, Hepatitis B, Human Immunodeficiency Virus (HIV), including hepatic disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 7 weeks
Incidence of Serious Adverse Events (SAEs) | up to 7 weeks
AEs leading to discontinuation | Up to 7 weeks
Number of clinically significant changes in vital signs | Up to 7 weeks
Number of clinically significant changes in ECG (electrocardiogram) | Up to 7 weeks
Number of clinically significant changes in physical examinations | Up to 7 weeks
Number of clinically significant changes in clinical laboratory tests | Up to 7 weeks

SECONDARY OUTCOMES:
Maximum observed concentration(Cmax)- Part A SAD | up to 7 weeks
Time of maximum observed concentration(Tmax)- Part A SAD | Up to 7 weeks
Terminal elimination rate constant (Lz)-Part A SAD | up to 7 weeks
Half life (T-HALF)- Part A SAD | Up to 7 weeks
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration(AUC(0-T)- Part A SAD | Up to 7 weeks
Area under the concentration-time curve from time zero extrapolated to infinite time(AUC(INF)-Part A SAD | Up to 7 weeks
Apparent total body clearance(CL/F)-Part A SAD | Up to 7 weeks
Apparent volume of distribution at terminal phase(Vz/F)- Part A SAD | Up to 7 weeks
Maximum observed concentration(Cmax)-Part B and Part C MAD | Up to 7 years
  For day 1 , day 13 and day 14
Time of maximum observed concentration(Tmax)-Part B and Part C MAD | Up tp 7 weeks
  For day 1, day 13 and day 14
Area under the concentration-time curve in one dosing interval(AUC(TAU)- Part B and Part C MAD | Up to 7 weeks
  For day 1 and day 14
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration(AUC(0-T)-Part B and Part C MAD | Up to 7 weeks
  For Day 14
Terminal elimination rate constant (Lz)-Part B and Part C MAD | up to 7 weeks
  For day 14
Half life (T-HALF)- Part B and Part C MAD | Up to 7 weeks
  For day 14
Apparent total body clearance(CL/F)-Part B and Part C MAD | Up to 7 weeks
  For day 14
Apparent volume of distribution at terminal phase(Vz/F)- Part B and Part C MAD | Up to 7 weeks
  For day 14
Accumulation Ratio Cmax (AR(Cmax)-Part B and Part C MAD | Up to 7 weeks
  For day 14
Accumulation Ratio AUC(TAU) (AR(AUC[TAU])- Part B and Part C MAD | Up to 7 weeks
  for day 14

CONTACTS AND LOCATIONS:
Locations (2):
- PRA Health Sciences - Groningen, Groningen, Netherlands
- Richmond Pharmacology, London, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm